CLINICAL TRIAL: NCT04507204
Title: Real-world Evidence of Duration of Adhansia XR for Treatment of ADHD (RE-DAX): An Open-label Pragmatic Study to Assess the Real-world Effectiveness of Adhansia XR in Treatment of Adult and Adolescent Patients With ADHD in the United States
Brief Title: Real-World Evidence of Duration of Effect of Adhansia XR (Extended-Release) for Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD)
Acronym: RE-DAX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: (due to administrative reasons not related to efficacy or safety.)
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADA4003
Record Dates: First submitted 2020-07-24; First posted 2020-08-11 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; Methylphenidate; Adhansia XR; MPH; OROS; Phase IV
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adhansia XR (Experimental): Adhansia XR capsules taken orally once daily with or without food.
  Interventions: Drug: Adhansia XR
- Concerta (Active Comparator): Concerta tablets taken orally once daily in the morning and swallowed whole with the aid of liquids, with or without food.
  Interventions: Drug: Concerta

INTERVENTIONS:
Drug: Adhansia XR — Methylphenidate extended-release capsules taken once daily (25 mg, 35 mg, 45 mg, 55 mg, 70 mg, and 85 mg)
  Other Names: Methylphenidate hydrochloride (HCl) extended release
  Arms: Adhansia XR
Drug: Concerta — An osmotic-controlled oral release delivery system (OROS) of methylphenidate HCl (MPH) extended-release tablets taken once daily (18 mg, 27 mg, 36 mg, and 54 mg)
  Other Names: Methylphenidate hydrochloride (HCl)
  Arms: Concerta

SUMMARY:
The purpose of this study is to investigate the treatment effectiveness of Adhansia XR at month-2 after initiation, and the effectiveness of Adhansia XR overall and when compared with the active comparator group (Concerta) over time.

DETAILED DESCRIPTION:
This phase IV study is a prospective, open-label, randomized, pragmatic study to investigate the treatment effectiveness of Adhansia XR at Month-2 after initiation, and the effectiveness of Adhansia XR overall and when compared with the active comparator group (OROS MPH or Concerta) over time. Additional outcome assessments for both treatment arms include Health-Related Quality of Life (HRQoL) during the 6-month follow-up period. The burden of illness (BOI) will be investigated by collecting additional measures such as healthcare resource utilization (HCRU), broader treatment patterns, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a physician-confirmed diagnosis of ADHD per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and the health care practitioner (HCP) has made the decision to prescribe an extended-release methylphenidate (ER MPH) product to the patient for potential improvement of symptoms throughout and later in the day, independent of this study.
* Patient must be 12 years of age or older.
* Patient must be eligible to receive Adhansia XR or osmotic- release oral delivery system methylphenidate ([OROS MPH] or Concerta) according to the US product labels; a patient must be eligible and willing to receive either drug, as randomization will assign them to a specific treatment group. Patient may be treatment-experienced or naïve to pharmacological therapy for ADHD, so long as all inclusion and no exclusion criteria are met.
* Patient must be willing to take only the assigned study medication per HCP instructions based on FDA label guidance for treatment of their ADHD for the first 2 months of the study (i.e. full titration period). Patients should not be on any other medication, or starting any new non-medication treatment, proven to have effect on ADHD in the first two months of the study.

Exclusion Criteria:

* Concurrent participation in an investigational study in which patient assessment and/or treatment may be dictated by a protocol.
* Patients with a true allergy to methylphenidate (MPH), amphetamine (AMP), or sympathomimetic amines, history of serious adverse reactions to MPH or AMP or be known to be non-responsive to MPH or AMP treatment.
* Patient is currently stable on their ADHD treatment regimen.
* Female patients of child bearing potential who are pregnant, planning on becoming pregnant or breastfeeding.
* Patient with any known conditions that are contraindicated for either Adhansia XR or OROS MPH (or Concerta) use, as documented in the US Full Prescribing Information, including patients with any known serious structural cardiac abnormalities, cardiomyopathy, serious heart arrhythmias, or coronary artery disease.
* Patients with a known sensitivity to the food dye tartrazine (Federal Food, Drug, and Cosmetic Yellow No. 5).
* Suicidal Ideation

  * The Columbia-Suicide Severity Rating Scale (C-SSRS) will be administered at screening and at Month-2, Month-4, and Month-6, but also depends on the judgment of the HCP.
* Inability or unwillingness of the patient (or parent/guardian if patient is a minor) to complete the study-required electronic questionnaires and provide required information through electronic means.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Harmonex, Inc., Dothan, Alabama
  - Southern California Research LLC, Beverly Hills, California
  - CT Clinical Research, Cromwell, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Eastern Research. Inc., Hialeah, Florida
  - Wellness Research Center Inc., Miami, Florida
  - AdventHealth Medical Group Pediatrics at Orange City, Orange City, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - Revive Research Institute, Elgin, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - BTC of New Bedford, LLC, New Bedford, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Mid-Ohio Behavioral Health, Columbus, Ohio
  - SFM Clinical Trials, Scotland, Pennsylvania
  - Rainbow Research, Barnwell, South Carolina
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Dixie Pediatrics, St. George, Utah
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Eastside Therapeutic Resource Inc dba Core Clinical Research, Everett, Washington
  - MultiCare Health System - Rockwood Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boesen K, Paludan-Muller AS, Gotzsche PC, Jorgensen KJ. Extended-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD012857. doi: 10.1002/14651858.CD012857.pub2. PMID 35201607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit was 30-Jul-2020; primary completion date was 22-Dec-2021 (i.e., the adult portion was completed). This study was statistically powered to conduct a separate analysis for adult and adolescent patients. However, enrollment of adolescents was unexpectedly slow as a result of the Coronavirus Disease 2019 (COVID-19) pandemic and a business decision was made on 31-Jan-2022 to discontinue enrollment of adolescents, thus terminating this branch of the study.
Groups:
- Adhansia XR: Methylphenidate extended-release capsules taken once daily.
Period: Overall Study
Arm/Group | Adhansia XR | Concerta
Started | 133 | 134
Completed | 83 | 86
Not Completed | 50 | 48
Not completed — Adverse Event | 8 | 13
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 15 | 14
Not completed — Poor Compliance with Protocol | 2 | 4
Not completed — Other (e.g., PI judgment, moved out of state. etc.) | 4 | 3
Not completed — Withdrawal of Patient Consent | 21 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adhansia XR | Concerta | Total
Number analyzed (Participants) | 133 | 134 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (11.7) | 38.6 (12.5) | 37.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 62 | 61 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 15 | 11 | 26
  White | 108 | 116 | 224
  Other | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 44
  Not Hispanic or Latino | 108 | 113 | 221
  Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD-Rating Scale 5 (ADHD-RS-5) Total Score From Baseline to Month 2 Among Patients Treated With Adhansia XR
Description: The ADHD-RS-5 assesses the frequency and severity of each of the 18 ADHD symptoms among adults based on DSM-5 criteria. Each of the 18 DSM-5 symptoms are rated on a 4 point scale from 0 (never or rarely) to 3 (very often), yielding a total score of 0 to 54. A higher score corresponds to worse ADHD severity.
Time Frame: Baseline to Month-2
Population: Full Analysis Set (FAS) Adult Population consisted of patients who were randomly assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adhansia XR
Number analyzed (Participants) | 133
score on a scale
  Total Score at baseline | 34.6 (8.60)
  Total Score at Month 2: number analyzed (Participants) | 99
  Total Score at Month 2 | 18.7 (9.01)

2. Secondary Outcome: Difference in Time Sensitive ADHD Symptom Scale (TASS) Between Treatment Groups to Establish Non-inferiority
Description: TASS was completed at the end of waking hours (14 - 16 hours post-dosing) at Month-2 after baseline visit. TASS was developed to capture the change in ADHD symptoms over the course of a day and consists of 18 items that directly correspond to the 18 ADHD symptom domains listed in the DSM-5. Each item is scored on a 4-point scale as follows: 0 (none), 1 (mild), 2 (moderate), and 3 (severe); the maximum total score is 54. A higher total score corresponds to worse ADHD severity.
Time Frame: Month-2
Population: FAS Adult Population consisted of patients who were randomly assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 105 | 122
score on a scale | 20.2 (0.93) | 22.1 (0.88)

3. Secondary Outcome: Assessment of Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S rates symptoms from 1 (not ill) to 7 (extremely ill). A higher score corresponds to higher ADHD severity.
Time Frame: Baseline, Month-2, Month-4, and Month-6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
score on a scale
  Baseline | 4.6 (0.08) | 4.6 (0.07)
  Month 2: number analyzed (Participants) | 99 | 107
  Month 2 | 3.1 (0.09) | 3.2 (0.08)
  Month 4: number analyzed (Participants) | 88 | 96
  Month 4 | 2.7 (0.09) | 3.0 (0.09)
  Month 6: number analyzed (Participants) | 94 | 99
  Month 6 | 2.7 (0.09) | 3.1 (0.09)

4. Secondary Outcome: Assessment of Clinical Global Impression-Improvement (CGI-I)
Description: The CGI-I measures global improvement prior to and after initiating the study medication. The CGI-I scale is 1 question, and rates improvement compared with the baseline visit using a 7-point scale. The range of responses are from 1 (very much improved) through 7 (very much worse). A higher score corresponds to higher ADHD severity.
Time Frame: Month-2, Month-4, and Month-6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 99 | 107
score on a scale
  Month 2 | 2.3 (0.10) | 2.3 (0.09)
  Month 4: number analyzed (Participants) | 88 | 96
  Month 4 | 2.0 (0.09) | 2.2 (0.09)
  Month 6: number analyzed (Participants) | 94 | 99
  Month 6 | 2.0 (0.11) | 2.3 (0.10)

5. Secondary Outcome: Assessment of Treatment Satisfaction
Description: The Treatment Satisfaction Questionnaire for Medications (TSQM) measures a patient's level of satisfaction or dissatisfaction with the study medication. It assesses perceptions of effectiveness, side effects and convenience of the medication and consists of 14 items that evaluate these three domains and one global scale item (ie, global satisfaction). Scores for each domain are computed by adding the TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100.
  A lower score indicates a lower satisfaction with treatment.
Time Frame: Month-1, Month-2, and Month-6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
score on a scale
  Global Satisfaction at Month 1: number analyzed (Participants) | 107 | 117
  Global Satisfaction at Month 1 | 84.8 (1.60) | 84.3 (1.55)
  Global Satisfaction at Month 2: number analyzed (Participants) | 92 | 92
  Global Satisfaction at Month 2 | 85.2 (1.83) | 82.8 (1.82)
  Global Satisfaction at Month 6: number analyzed (Participants) | 70 | 75
  Global Satisfaction at Month 6 | 86.2 (1.98) | 84.3 (1.92)
  Effectiveness at Month 1: number analyzed (Participants) | 107 | 117
  Effectiveness at Month 1 | 51.3 (1.91) | 52.4 (1.84)
  Effectiveness at Month 2: number analyzed (Participants) | 92 | 92
  Effectiveness at Month 2 | 61.1 (1.94) | 58.8 (1.92)
  Effectiveness at Month 6: number analyzed (Participants) | 70 | 75
  Effectiveness at Month 6 | 63.9 (2.69) | 61.9 (2.61)
  Side Effects at Month 1: number analyzed (Participants) | 107 | 117
  Side Effects at Month 1 | 74.0 (2.93) | 69.6 (2.82)
  Side Effects at Month 2: number analyzed (Participants) | 92 | 92
  Side Effects at Month 2 | 72.0 (3.26) | 67.6 (3.24)
  Side Effects at Month 6: number analyzed (Participants) | 70 | 75
  Side Effects at Month 6 | 70.7 (3.48) | 74.1 (3.37)
  Convenience at Month 1: number analyzed (Participants) | 47 | 60
  Convenience at Month 1 | 58.9 (1.81) | 59.2 (1.63)
  Convenience at Month 2: number analyzed (Participants) | 42 | 48
  Convenience at Month 2 | 57.0 (1.90) | 58.7 (1.78)
  Convenience at Month 6: number analyzed (Participants) | 35 | 32
  Convenience at Month 6 | 59.7 (2.10) | 57.0 (2.13)

6. Secondary Outcome: Healthcare Resource Utilization (HCRU)
Description: A comparison of the frequency of health care encounters between the 2 treatment groups. Healthcare resource utilization were evaluated monthly by comparing the frequency of clinic visits (outpatient), inpatient/hospitalizations (and length of stay), and emergency department visits between the 2 treatment groups.
Time Frame: Baseline (past 6 months) Months -2, -4, and -6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Visits or Inpatient Admissions
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
Visits or Inpatient Admissions
  Baseline (past 6 months) Overall Total Visits or Inpatient Admissions | 2.14 (0.314) | 2.93 (0.314)
  Month 2 - Overall Total Visits or Inpatient Admissions: number analyzed (Participants) | 99 | 108
  Month 2 - Overall Total Visits or Inpatient Admissions | 2.26 (0.542) | 2.43 (0.481)
  Month 4 - Overall Total Visits or Inpatient Admissions: number analyzed (Participants) | 88 | 96
  Month 4 - Overall Total Visits or Inpatient Admissions | 1.67 (0.474) | 1.73 (0.504)
  Month 6 - Overall Total Visits or Inpatient Admissions: number analyzed (Participants) | 95 | 99
  Month 6 - Overall Total Visits or Inpatient Admissions | 1.34 (0.515) | 1.85 (0.480)

7. Secondary Outcome: Adult ADHD Quality of Life Scale - Revised (AAQoL-R)
Description: Used to assess health-related quality of life for adult patients. The AAQoL yields a total score based on 29 items. The raw scores are transformed to a 0 to 100 scale with higher scores indicating a better quality of life.
Time Frame: Baseline, Months -1, -2, -3, -4, -5 and -6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
score on a scale
  Total Score at Baseline: number analyzed (Participants) | 122 | 129
  Total Score at Baseline | 41.1 (1.19) | 41.1 (1.16)
  Total Score at Month 1: number analyzed (Participants) | 111 | 120
  Total Score at Month 1 | 55.5 (1.24) | 55.0 (1.20)
  Total Score at Month 2: number analyzed (Participants) | 96 | 97
  Total Score at Month 2 | 63.0 (1.31) | 59.1 (1.29)
  Total Score at Month 3: number analyzed (Participants) | 88 | 99
  Total Score at Month 3 | 63.4 (1.38) | 60.9 (1.30)
  Total Score at Month 4: number analyzed (Participants) | 81 | 90
  Total Score at Month 4 | 64.7 (1.43) | 61.8 (1.36)
  Total Score at Month 5: number analyzed (Participants) | 83 | 88
  Total Score at Month 5 | 66.3 (1.44) | 60.2 (1.39)
  Total Score at Month 6: number analyzed (Participants) | 72 | 77
  Total Score at Month 6 | 67.4 (1.52) | 63.6 (1.48)

8. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: The WPAI questionnaire is designed to measure the effect of general health and symptom severity on work productivity and regular activities during the past 7 days. It consists of 4 domains [absenteeism (missing work), presenteeism (impaired productivity at work), overall work performance (combined absenteeism and presenteeism), and non-work activities (activity impairment)]. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Months -2, -3, -4, -5, and -6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of impairment
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
percentage of impairment
  Percent work time missed due to health (Absenteeism) - Baseline: number analyzed (Participants) | 88 | 85
  Percent work time missed due to health (Absenteeism) - Baseline | 5.4 (1.26) | 5.6 (1.28)
  Percent work time missed due to health (Absenteeism) - Month 2: number analyzed (Participants) | 72 | 63
  Percent work time missed due to health (Absenteeism) - Month 2 | 4.2 (1.48) | 3.7 (1.64)
  Percent work time missed due to health (Absenteeism) - Month 3: number analyzed (Participants) | 70 | 67
  Percent work time missed due to health (Absenteeism) - Month 3 | 3.0 (1.57) | 3.2 (1.62)
  Percent work time missed due to health (Absenteeism) - Month 4: number analyzed (Participants) | 62 | 61
  Percent work time missed due to health (Absenteeism) - Month 4 | 2.4 (1.61) | 4.7 (1.72)
  Percent work time missed due to health (Absenteeism) - Month 5: number analyzed (Participants) | 63 | 62
  Percent work time missed due to health (Absenteeism) - Month 5 | 4.8 (1.62) | 4.9 (1.70)
  Percent work time missed due to health (Absenteeism) - Month 6: number analyzed (Participants) | 55 | 57
  Percent work time missed due to health (Absenteeism) - Month 6 | 2.9 (1.72) | 4.1 (1.82)
  Percent impairment while working due to health (Presenteeism) - Baseline: number analyzed (Participants) | 86 | 85
  Percent impairment while working due to health (Presenteeism) - Baseline | 32.0 (2.16) | 33.3 (2.18)
  Percent impairment while working due to health (Presenteeism) - Month 2: number analyzed (Participants) | 72 | 64
  Percent impairment while working due to health (Presenteeism) - Month 2 | 19.7 (2.52) | 24.2 (2.69)
  Percent impairment while working due to health (Presenteeism) - Month 3: number analyzed (Participants) | 66 | 66
  Percent impairment while working due to health (Presenteeism) - Month 3 | 20.1 (2.73) | 25.0 (2.70)
  Percent impairment while working due to health (Presenteeism) - Month 4: number analyzed (Participants) | 59 | 56
  Percent impairment while working due to health (Presenteeism) - Month 4 | 13.5 (2.75) | 24.6 (2.91)
  Percent impairment while working due to health (Presenteeism) - Month 5: number analyzed (Participants) | 63 | 60
  Percent impairment while working due to health (Presenteeism) - Month 5 | 17.8 (2.76) | 18.3 (2.90)
  Percent impairment while working due to health (Presenteeism) - Month 6: number analyzed (Participants) | 55 | 54
  Percent impairment while working due to health (Presenteeism) - Month 6 | 15.9 (2.91) | 17.6 (3.14)
  Percent overall work impairment due to health - Baseline: number analyzed (Participants) | 85 | 83
  Percent overall work impairment due to health - Baseline | 34.1 (2.31) | 35.5 (2.34)
  Percent overall work impairment due to health - Month 2: number analyzed (Participants) | 71 | 62
  Percent overall work impairment due to health - Month 2 | 22.4 (2.71) | 27.2 (2.93)
  Percent overall work impairment due to health - Month 3: number analyzed (Participants) | 64 | 65
  Percent overall work impairment due to health - Month 3 | 21.8 (2.94) | 26.4 (2.94)
  Percent overall work impairment due to health - Month 4: number analyzed (Participants) | 58 | 56
  Percent overall work impairment due to health - Month 4 | 15.8 (2.94) | 25.3 (3.16)
  Percent overall work impairment due to health - Month 5: number analyzed (Participants) | 62 | 59
  Percent overall work impairment due to health - Month 5 | 19.7 (2.98) | 19.5 (3.17)
  Percent overall work impairment due to health - Month 6: number analyzed (Participants) | 54 | 54
  Percent overall work impairment due to health - Month 6 | 18.4 (3.15) | 18.9 (3.37)
  Percent activity impairment due to health - Baseline: number analyzed (Participants) | 117 | 126
  Percent activity impairment due to health - Baseline | 39.7 (2.05) | 40.9 (1.98)
  Percent activity impairment due to health - Month 2: number analyzed (Participants) | 92 | 92
  Percent activity impairment due to health - Month 2 | 26.1 (2.33) | 30.1 (2.30)
  Percent activity impairment due to health - Month 3: number analyzed (Participants) | 86 | 97
  Percent activity impairment due to health - Month 3 | 26.1 (2.44) | 27.1 (2.29)
  Percent activity impairment due to health - Month 4: number analyzed (Participants) | 79 | 84
  Percent activity impairment due to health - Month 4 | 19.5 (2.52) | 28.6 (2.45)
  Percent activity impairment due to health - Month 5: number analyzed (Participants) | 81 | 87
  Percent activity impairment due to health - Month 5 | 23.6 (2.54) | 26.3 (2.43)
  Percent activity impairment due to health - Month 6: number analyzed (Participants) | 69 | 76
  Percent activity impairment due to health - Month 6 | 21.9 (2.72) | 23.5 (2.60)

9. Secondary Outcome: Patient Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is an instrument used to measure the quality and patterns of sleep; It differentiates "poor" from "good" sleep. It is filled out by the caregiver or the patient and the global sum score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Time Frame: Baseline and Months -2, -4, and -6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adhansia XR | Concerta
Number analyzed (Participants) | 133 | 134
score on a scale
  Global PSQI - Baseline: number analyzed (Participants) | 118 | 129
  Global PSQI - Baseline | 9.68 (0.219) | 9.59 (0.209)
  Global PSQI - Month 2: number analyzed (Participants) | 93 | 95
  Global PSQI - Month 2 | 7.92 (0.251) | 9.59 (0.209)
  Global PSQI - Month 4: number analyzed (Participants) | 79 | 89
  Global PSQI - Month 4 | 8.11 (0.268) | 7.76 (0.252)
  Global PSQI - Month 6: number analyzed (Participants) | 71 | 75
  Global PSQI - Month 6 | 7.92 (0.284) | 7.80 (0.273)

ADVERSE EVENTS:
Time Frame: All adverse events were reported starting from the time informed consent for study participation up to 6 months.
Description: Since participants may have received multiple dose levels during the study and a participant may have experienced an adverse event which started on one dose level and was ongoing at subsequent dose level(s), the adverse events are presented for all dose levels combined.
Arm/Group | Adhansia XR | Concerta
All-Cause Mortality (participants affected / at risk) | 0/133 | 1/134
Serious Adverse Events (participants affected / at risk) | 3/133 | 4/134
Other Adverse Events (participants affected / at risk) | 28/133 | 27/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adhansia XR (N=133) | Concerta (N=134)
Delusion (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 3
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adhansia XR (N=133) | Concerta (N=134)
Decreased appetite (Metabolism and nutrition disorders) | 10 | 10
Anxiety (Psychiatric disorders) | 5 | 11
Insomnia (Psychiatric disorders) | 13 | 5
Headache (Nervous system disorders) | 4 | 7
Dry Mouth (Gastrointestinal disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04507204/Prot_SAP_002.pdf